CLINICAL TRIAL: NCT04670276
Title: Conservative Treatment of Gastrointestinal Fistulas by Endoscopic Injection of Emulsified Adipose Tissue Stromal Vascular Fraction (tSVFem)
Brief Title: Conservative Treatment of Gastrointestinal Fistulas by Endoscopic Injection of tSVFem
Acronym: tSVFem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Venanzio Porziella, Assistant professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3127 prot.num 0043082/20
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Fistula
Keywords: gastrointestinal fistula; Adipose-derived stem cells; adipose tissue stromal vascular fraction; Endoscopy
MeSH Terms: conditions — Digestive System Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients treated by endoscopic injection of emulsified adipose tissue stromal vascular fraction
  Interventions: Procedure: injection of emulsified adipose tissue stromal vascular fraction

INTERVENTIONS:
Procedure: injection of emulsified adipose tissue stromal vascular fraction — Endoscopic injection of 10 cc of autologous microfat into the fistula (through a 6-French catheter), until it was completely filled, and a total of 1-2 cc of tSVFem (through a 22G endoscopic needle) into the submucosa of the 4 quadrants of the fistula borders, to obliterate it completely.

SUMMARY:
Gastrointestinal (GI) fistula is a complex condition with high mortality and requiring a multidisciplinary management.

The aim of this study is to exploit the regenerative-tissue capacities of autologous emulsified adipose tissue-derived stromal vascular fraction (tSVFem, widely used in other medical fields - like plastic surgery -for different purposes) harvested and delivered locally by endoscopy to close the GI fistula.

The proposed technique for the treatment of GI fistulas with tSVFem requires a minimal, inexpensive, easily reproducible mechanical manipulation of autologous adipose tissue without necessity of any enzymatic digestion or cell expansion.

DETAILED DESCRIPTION:
Gastrointestinal fistula may be a life-threatening condition caused by several types of injuries (iatrogenic, traumatic, post-operative), requiring complex and multidisciplinary management. To date, no clear guidelines have been drawn up for the treatment, that may include a conservative, minimally invasive, or major surgical approach depending on the patient's specific clinical characteristics. Furthermore, patients with fistulas are often fragile, and surgical treatments are highly risky and invasive. Less invasive treatments such as stenting, endoluminal endoscopic vacuum therapy and suturing are widely employed, but these treatments often require long hospitalization, highly skilled operators, without certain results and with high rates of complications.

The aim of this study is to exploit the regenerative-tissue capacities of autologous emulsified adipose tissue-derived stromal vascular fraction (tSVFem, widely used in other medical fields - like plastic surgery -for different purposes) harvested and delivered locally by endoscopy to close the GI fistula. Indeed, the anti-inflammatory and regenerative-tissue promoting effects of tSVFem may safely promote rapid and effective tissue healing as alternative, and in this setting they were not investigated before. Fistulas are often long-standing chronic conditions, thus healing mechanisms are delayed and subverted in favor of inflammation and fibrosis, resembling chronic inflammatory diseases. Delivery of tSVFem is a promising new approach that promotes healing in virtue of its immunosuppressive, immunomodulatory, pro-angiogenic and regenerative potentials. Since the grafted material used in this study is autologous, there is no risk for rejection. All the procedures are performed under general anesthesia with orotracheal intubation or laryngeal mask. Approximately 30 cc of fat are harvested from the superficial layer of subcutaneous tissue by a 2.1 mm microcannula with 4, 1-mm size holes, arranged in a single raw, to get the so-called "microfat". Twenty cc of the harvested microfat are mechanical emulsified by sequential passages through 2.4mm and 1.2mm filters, and a 600/400 μm disposable filtering device.

Then the material is centrifuged at 3000 rounds for three minutes, obtaining the tSVFem after removal of supernatant fraction and oil released upon mature adipocytes mechanical disruption.

Subsequently, an endoscopy is performed to inject 10 cc of microfat into the fistula (through a 6-French catheter) until it was completely filled. Then, with a 22 Gauge endoscopic needle, a total of 1-2 cc of tSVFem were injected into the submucosa of the 4 quadrants of the fistula borders, to obliterate it completely.

A radiologic and endoscopic control at day-7 is done to evaluate complete healing of the fistula.

The technique proposed by the investigators for the treatment of GI fistulas with tSVFem requires a minimal, inexpensive, easily reproducible mechanical manipulation of autologous adipose tissue without necessity of any enzymatic digestion or cell expansion.

ELIGIBILITY:
Inclusion criteria:

• Patients affected by GI fistulas, not fit for surgical treatments of after failure of conventional conservative treatments

Exclusion Criteria:

* Enteroenteric fistulas
* Patients who do not sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-03-02 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Fistula healing | 7 days after the injection procedure of tSVFem
  Rate of healing of fistula at endoscopy and gastrografin swallow

SECONDARY OUTCOMES:
Incidence of treatment adverse events and complications | During the procedure, 7 days after and at 1-2 month follow-up
  To evaluate the percentage of patients that developed adverse events or any complications during and after the treatment proposed

CONTACTS AND LOCATIONS:
Overall Officials: Venanzio Porziella, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brinster CJ, Singhal S, Lee L, Marshall MB, Kaiser LR, Kucharczuk JC. Evolving options in the management of esophageal perforation. Ann Thorac Surg. 2004 Apr;77(4):1475-83. doi: 10.1016/j.athoracsur.2003.08.037. PMID 15063302
- [Background] Porziella V, Nachira D, Boskoski I, Trivisonno A, Costamagna G, Margaritora S. Emulsified stromal vascular fraction tissue grafting: a new frontier in the treatment of esophageal fistulas. Gastrointest Endosc. 2020 Dec;92(6):1262-1263. doi: 10.1016/j.gie.2020.06.019. Epub 2020 Jul 4. No abstract available. PMID 32634381
- [Background] Kuehn F, Loske G, Schiffmann L, Gock M, Klar E. Endoscopic vacuum therapy for various defects of the upper gastrointestinal tract. Surg Endosc. 2017 Sep;31(9):3449-3458. doi: 10.1007/s00464-016-5404-x. Epub 2017 Jan 11. PMID 28078463
- [Background] Brangewitz M, Voigtlander T, Helfritz FA, Lankisch TO, Winkler M, Klempnauer J, Manns MP, Schneider AS, Wedemeyer J. Endoscopic closure of esophageal intrathoracic leaks: stent versus endoscopic vacuum-assisted closure, a retrospective analysis. Endoscopy. 2013 Jun;45(6):433-8. doi: 10.1055/s-0032-1326435. Epub 2013 Jun 3. PMID 23733727
- [Background] Ceccarelli S, Pontecorvi P, Anastasiadou E, Napoli C, Marchese C. Immunomodulatory Effect of Adipose-Derived Stem Cells: The Cutting Edge of Clinical Application. Front Cell Dev Biol. 2020 Apr 17;8:236. doi: 10.3389/fcell.2020.00236. eCollection 2020. PMID 32363193
- [Background] Angelo Trivisonno, Marc Abecassis, Massimo Monti et al. Adipose Tissue: From Energy Reservoir to a Source of Cells for Epithelial Tissue Engineering. In: Stem Cells in Aesthetic Procedures: Springer Berlin Heidelberg,2014:303-326
- [Background] Trivisonno A, Nachira D, Boskoski I, Calcagni F, Tringali A, Costamagna G, Margaritora S, Porziella V. Autologous Fat Grafting Restores Soft-tissue Contour Deformities after Vascular Anomaly: Widening the Horizons of Employment of Autologous Fat Grafting. Plast Reconstr Surg Glob Open. 2019 Nov 27;7(11):e2518. doi: 10.1097/GOX.0000000000002518. eCollection 2019 Nov. No abstract available. PMID 31942308
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896